CLINICAL TRIAL: NCT05417932
Title: A Phase 1/ 2a, Multicenter Study of SCG101 in the Treatment of Subjects With Hepatitis B Virus-Related Hepatocellular Carcinoma
Brief Title: A Study of SCG101 in the Treatment of Subjects With Hepatitis B Virus-Related Hepatocellular Carcinoma
Acronym: TCR-T
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SCG Cell Therapy Pte. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCG101-UR-103
Record Dates: First submitted 2022-05-24; First posted 2022-06-14 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Hepatitis B Virus Related Hepatocellular Carcinoma; Hepatocellular Carcinoma Recurrent
Keywords: HCC; Hepatitis B Virus Related; HCC Recurrent

STUDY DESIGN:
Intervention Model Description: SCG101 in the Treatment of Subjects with Hepatitis B Virus-Related Hepatocellular Carcinoma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SCG101 (Experimental): This is a single arm study.
  Patients will receive infusion and will be observed for dose limiting toxicity (DLT) over a 28-day period, and thereafter enter the progression free survival observation period and continuous long term survival follow up at time of disease progression.
  Interventions: Biological: SCG101

INTERVENTIONS:
Biological: SCG101 — Infusion of HBsAg-specific TCR autologous T cells at assigned dose levels.

SUMMARY:
This Phase 1/ 2a study is a multicenter study to evaluate the safety, tolerability and efficacy of SCG101 in subjects with hepatitis B virus-related hepatocellular carcinoma

DETAILED DESCRIPTION:
This study will be conducted in 2 parts: In Phase 1 dose escalation, cohorts of 3-6 subjects each will be sequentially assigned to escalating dose level of SCG101. The recommended phase 2 dose (RP2D) will be selected based on the safety, PK/ PD and antitumor activities if the maximum tolerated dose (MTD) is not reached from the planned dose levels.

In Phase 2a, subjects will be enrolled to characterize the safety and evaluate the efficacy of SCG101.

ELIGIBILITY:
Main Inclusion Criteria:

* Histologically or cytologically confirmed Hepatocellular carcinoma (HCC)
* Subjects with HCC who have received at least 2 standard systemic therapies
* HLA-A *02
* BCLC stage B or C
* Child-pugh score ≤ 7
* Serum HBeAg negative, serum (or tumor tissue) HBsAg positive, and serum HBV-DNA must be 2 × 1000 IU/ml
* Have at least one measurable leasion at baseline as per mRECIST and RECIST v1.1 criteria
* Life expectancy of 3 months or greater
* Ability to provide informed consent form
* Ability to comply with all the study procedures

Main Exclusion Criteria:

* Subjects with history of another primary cancer
* Untreated or active central nervous system (CNS) or leptomeningeal metastasis, or history of hepatic encephalopathy, or other clinically significant CNS diseases
* Autoimmune diseases requiring immunosuppressive therapy (except topical medication) or subjects with significant persistent immune rejection
* Known history of neurological or mental disorder, including epilepsy or dementia
* Known history of positive results for human immunodeficiency virus (HIV) 1 or 2 or known acquired immunodeficiency syndrome (AIDS)
* Prior exposure to any cell therapy such as, but not limited to killer (NK) cells, cytokine-induced killer (CIK) cells, dendritic cells (DC), cytotoxic T lymphocytes (CTL), stem cell therapy, CAR T/TCR T cell therapy
* Allergy to immunotherapy drugs and lymphodepleting chemotherapy (cyclophosphamide and fludarabine)
* Any subjects who cannot be evaluated by either triphasic liver CT or triphasic MRI because of allergy or other contraindication to both CT and MRI contrast agents
* Any condition which, in the investigator's opinion, makes the subject unsuitable for trial participation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2022-10-26 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of SCG101 | Start of SCG101 infusion until 100 days post SCG101 infusion
  Based on incidence of adverse events (AE) using NCI-CTCAE v5.0
Tumor response of SCG101 (Phase 2) | Start of SCG101 infusion until a complate response or partial response is observed, disease progression, and long term survival follow up up to 15 years

SECONDARY OUTCOMES:
Preliminary clinical efficacy of SCG101 | Start of SCG101 infusion until a complete response or partial response is observed after 28 days from SCG101 infusion.
  Objective response rate
Antiviral activity before and after SCG101 infusion | Start of SCG101 infusion and throughout DLT and PFS until disease progression, an average of 24 months.
  Based on changes in serum levels of HBsAg
Change in pharmacodynamic markers (PD) before and after SCG101 infusion | Start of SCG101 infusion and throughout DLT and PFS until disease progression, an average of 24 months.
  Based on changes in serum from the liver function
Persistence of viral vector copy number (VCN) after SCG101 infusion | Start of SCG101 infusion until disease progression, an average of 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: SCG Cell Therapeutics, Study Director — SCG Cell Therapy Pte. Ltd.
Locations (4):
- New York, New York, New York, United States
- Hong Kong (2):
  - Hong Kong is., Hong Kong
  - Hong Kong NT, Hong Kong
- Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No